CLINICAL TRIAL: NCT01368159
Title: Randomised, Comparative Trial in Parallel Groups and Blinded, to Compare Efficacy on Pain Following a Procedure for Injecting Sclerotherapeutic Foam Into the G.S V. Under Echography Control, Between Three Types of Medical Compression Hose
Brief Title: Efficacy on Pain Following a Procedure for Injecting Sclerotherapeutic Foam Into the Great Saphenous Vein
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Le Club Mousse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Classmousse1
Record Dates: First submitted 2011-04-13; First posted 2011-06-07 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Venous Disease
MeSH Terms: interventions — Stockings, Compression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- pressure centred at 25 mm Hg (Active Comparator)
  Interventions: Device: Compression Stockings
- pressure between 20 and 36 mm Hg (Active Comparator)
  Interventions: Device: Compression Stockings
- pressure between 10 and 15 mm Hg (Placebo Comparator)
  Interventions: Device: Compression Stockings

INTERVENTIONS:
Device: Compression Stockings — The trial objectives are to compare efficacy relative to pain, along the route of the vein following echoguided endovenous injection of sclerotherapeutic foam into the Great Saphenous vein, of class III microfibre compression (centred at 25 mm Hg) versus class I (10-15 mm Hg) versus class III cotton compression (20 to 36 mm Hg) over 21 days. The main contrast will be the comparison between the first two groups mentioned. All other contrasts will be secondary. The "Class I compression" versus "The two class III compressions" contrast will also be studied.
  Other Names: ACTYS 25 ®; Varisma Comfort Coton ®; Varisma Séduction ®

SUMMARY:
The trial objectives are to compare efficacy relative to pain, along the route of the vein following echoguided endovenous injection of sclerotherapeutic foam into the Great Saphenous vein, of class III microfibre compression (centred at 25 mm Hg) versus class I (10-15 mm Hg) versus class III cotton compression (20 to 36 mm Hg) over 21 days. The main contrast will be the comparison between the first two groups mentioned. All other contrasts will be secondary. The "Class I compression" versus "The two class III compressions" contrast will also be studied.

Efficacy will be measured by totalling the VAS scores for maximum pain experienced since the morning and evaluated by the patient at the end of the day.

Consumption of analgesics or the number of days of analgesic treatment necessary for the 3 compression types used will be compared.

One of the trial objectives is also to show that regular use of a class III compression product leads to a reduction in complications following sclerosis (by reducing the number of non-serious/serious complications specific to sclerosis: matting, pigmentation, inflammation, development of sclerosis requiring drainage, DVT, pulmonary embolism, etc.). The trial also aims to compare the rate of successful sclerosis between the three devices, success being defined by complete or partial occlusion of the great saphenous vein, leading to the disappearance of reflux at the crural level.

The other secondary objectives will be patient evaluation of comfort, ease of putting on and taking off the compression hose and a global appreciation of the procedure for echoguided endovenous injection of sclerotherapeutic foam into the great saphenous vein, followed by wearing compression hose.

DETAILED DESCRIPTION:
Not desired

ELIGIBILITY:
Inclusion Criteria:

General:

* Patient at least 18 years old
* Patient agreeing to give her informed consent in writing
* Patient taking effective contraceptive on inclusion and not planning pregnancy during the trial period.
* Patient registered with the social security or equivalent regime;

Linked to the pathology:

* Patient suffering from truncal insufficiency of the SVG supplied either by reflux from the saphenofemoral junction, with or without competent terminal valve, or by collaterals or perineal varicosities in the subinguinal region and who is scheduled to have endovenous injection of sclerotherapeutic foam into the great saphenous vein presenting truncal reflux of at least one second, the diameter of which is at least 4 mm (no limit for maximum calibre) standing 15 cm from the inguinal fold (according to an echo-doppler taken less than three months prior to inclusion).
* Injection initially planned of 2% Aetoxisclerol, the injection volume of which is limited to 3 ml of liquid, i.e. less than 15 ml of foam, for complete filling of the great saphenous and a spasm. (to standardise the procedure before fitting the compression hose) Patient classified C2 to C5 (clinical stages in CEAP classification).

Exclusion Criteria:

* General:
* Patient regularly taking analgesics or anti-inflammatories.
* Patient suffering from a state or prior history of mental or psychiatric disorder or any other factor limiting aptitude to take an informed part and respect of the protocol; Patient suffering from chronic hepatopathology.
* Renal insufficiency (clearance < 60 ml/min. according to Cockcroft).
* Patient suffering from a known evolving malignant pathology.
* Patient suffering from decompensated cardiac or respiratory insufficiency.
* Patient who is pregnant or breast-feeding.
* Patient currently taking part in a clinical trial or who took part in a clinical trial during the month preceding inclusion.
* Person deprived of liberty by a legal or administrative decision, Adult patient protected by the law, under legal protection or guardianship.

Linked to the pathology/product:

* Patient suffering from LL pain other than vascular (sciatica, gonarthrosis, neuropathy, etc.)
* Patient presenting contraindications for class III venous compression (20 to 36 mmHg)
* Patient with a prior history of skin reactions following the use of venous compression products
* Scheduling a procedure for endovenous injection other than into the great saphenous vein during the period of study of the leg, planned during the 2 months following SVG sclerosis.
* Patient displaying post-thrombotic or primary anomalies of the deep vein network on the Echo-Doppler (less than 3 months before inclusion).
* Patient suffering from arteriopathy of the lower limbs with a systolic pressure index at the ankle of < 0.6
* Saphenous incompetence not meeting the anatomical and/or haemodynamic criteria defined in the inclusion criteria.
* Open ulcer in the LL (C6 of CEAP classification).
* Patient not tolerating compression or requiring chronic fitting of high pressure compression (in excess of 20 mmHg).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
pain following a procedure for injecting sclerotherapeutic foam into the Great Saphenous vein under echography control | 25 days
  Pain evaluated from D1 to D21 by the patient at the end of the day using a vertical visual analog scale (VAS) on 10 cm not fixed, in the patient's book: "Indicate the maximum intensity of your pain along the route of the treated vein since this morning and before taking any analgesic. Draw a horizontal line on the vertical line below

CONTACTS AND LOCATIONS:
Overall Officials: Charles ZARCA, MD, Principal Investigator — Le Club Mousse